CLINICAL TRIAL: NCT06818201
Title: Effects of Transcranial Direct Current Stimulation Over Motor Cortex During Recovery of ACL Patients
Brief Title: Effects of tDCS on Motor Cortex During ACL Recovery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Universidad Católica de Valencia San Vicente Mártir (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UCV/2023-2024/053
Record Dates: First submitted 2025-01-24; First posted 2025-02-10 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-01

CONDITIONS: Anterior Cruciate Ligament Reconstruction Rehabilitation
Keywords: motor control; Anterior Cruciate Ligament; exercise; tDCS
MeSH Terms: conditions — Motor Activity | interventions — Rehabilitation

STUDY DESIGN:
Intervention Model Description: To evaluate the effects of combined tDCS and exercise-based rehabilitation targeting neuromuscular control, comparing it to sham tDCS treatment.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The groups will be randomly assigned, and a double-blind procedure will be employed as the masking technique. Subject selection will be conducted randomly using the EPIDAT 3.1 program. Both the participants and the researcher responsible for data collection will remain unaware of the assigned intervention and the results obtained, respectively, until the study's conclusion. An independent researcher will generate a table of random numbers using an Excel formula to blind data collectors and outcome adjudicators, thereby ensuring unbiased outcome ascertainment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NIBS + rehabilitation (Experimental): The intervention using tDCS will be performed through the Home tDCS device (Ionclinics®). It will be introduced in the first part of the rehabilitation, during activation, because the required exercises will be of lower intensity, complexity, and more compatible with this intervention.
  Interventions: Device: NIBS; Procedure: Rehabilitation
- ShamNIBS + RHB (Sham Comparator): The device will be configured to produce an ascending ramp lasting 30 seconds, identical to the one used in the experimental group, followed by a descending ramp of another 30 seconds. Thus, the control group will experience a sensation of tingling on the scalp, similar to that felt by the experimental group. This stimulation will have a total duration of 1 minute, which will not be sufficient to induce changes in cortical excitability
  Interventions: Procedure: Rehabilitation; Behavioral: Sham Comparator

INTERVENTIONS:
Device: NIBS — A total of 16 sessions will be scheduled, distributed over 8 weeks (2 sessions/week). The continuous current intensity will be set at 2 mA, for 20 minutes. Two electrodes, anode (red) and cathode (black), will be used along with two sponge pads with conductive gel, all combined into a helmet for each patient. The electrodes will be placed according to the international 10-20 system in tDCS. The stimulated area will be the primary motor cortex (M1), so the anode will be placed at the C3 or C4 points and the cathode will be placed at the contralateral supraorbital area Fp1 or Fp2.
  Arms: NIBS + rehabilitation
Procedure: Rehabilitation — This protocol will consist of 72 sessions, distributed as 3 sessions per week over a period of 24 weeks. Strength will be the prioritized method of work and will be present in all phases. Additionally, periodic measurements will be included to ensure that the patient is making adequate progress and meets the necessary progression criteria to advance to the next phase
Behavioral: Sham Comparator — The device will be configured to produce an ascending ramp lasting 30 seconds, identical to the one used in the experimental group, followed by a descending ramp of another 30 seconds. Thus, the control group will experience a sensation of tingling on the scalp, similar to that felt by the experimental group. This stimulation will have a total duration of 1 minute, which will not be sufficient to induce changes in cortical excitability
  Arms: ShamNIBS + RHB

SUMMARY:
Anterior Cruciate Ligament (ACL) is a prevalent injury, particularly among young and physically active individuals. The efficacy of transcranial direct current stimulation (tDCS) and exercise-based rehabilitation on neuromuscular control in post-ACL reconstruction patients is evaluated, and these techniques are combined.

DETAILED DESCRIPTION:
Anterior cruciate ligament (ACL) rupture is a common injury, particularly among young and physically active individuals, with an incidence of 0.4 to 0.8 injuries per 1,000 person-years. While the majority of ruptures occur during sports activities (65-75%), a significant proportion (25-35%) happen in non-sport settings. Rehabilitation is crucial for recovery, but only 65% of patients return to their pre-injury activity level, and only 55% resume competitive activities. Neuromuscular structures such as the hamstrings and hip abductors play a vital role in reducing the risk of re-injury and aiding post-surgical rehabilitation.

Arthrogenic muscle inhibition (AMI) is a common phenomenon following ACL surgery, affecting quadriceps activation and force generation. While spinal mechanisms of AMI have been extensively studied, the influence of supraspinal centers, such as the motor cortex, in modulating AMI is also recognized. Traditional treatments, such as electrostimulation, are largely ineffective, and non-invasive brain stimulation techniques, such as transcranial direct current stimulation (tDCS), combined with exercise rehabilitation, are being explored to improve neuromuscular control.

This study aims to evaluate the effects of combined tDCS and exercise-based rehabilitation, comparing it to sham tDCS treatment. Outcomes will include cortical reorganization, corticospinal activation, pain perception, and psychosocial and functional variables. The central hypothesis is that reducing cortical hyperexcitability will enhance neuromuscular control, leading to improved outcomes and a reduced risk of re-injury.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis complete ACL tear through clinical evaluation and MRI imaging.
* Patients who have received surgical intervention.
* Aged between 16 and 40 years.
* Tegner activity level of 4 or higher.

Exclusion Criteria:

* Rupture, such as tendons, cartilage, bones, or ligaments.
* Absence of any pre-existing or current lower limb pathologies, such as open surgeries, knee arthroscopies, or femur/tibia fractures.
* Neuromuscular or metabolic diseases.
* Concussion within the past six months are not eligible.
* Cranial surgery or have intracranial metal clips are ineligible.
* Taking medications that affect neuronal activity.
* Neurological diseases or disorders are not eligible for participation.

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-11-28 (Actual); Primary Completion 2027-12-27 (Estimated); Study Completion 2027-12-27 (Estimated)

PRIMARY OUTCOMES:
Electromyography (EMGs) | At baseline, 90days post-surgery, 180days post-surgery
  The The Surface EMG amplitudes of the quadriceps and hamstring muscles. The main device, Musclelab, is equipped with a Musclelab force sensor and wireless surface elec-tromyography (EMGs). Electrode placement will follow the Surface ElectroMyoGraphy for the Non-Invasive Assessment of Muscle (SENIAM) protocol from the European Concerted Action in the Biomedical Health and Research Program (BIOMED II). The instructions provided to the patients will be to perform the movement with the max-imum possible contraction, and as rapidly as possible, to achieve the highest peak of force. The patient will carry out 3 familiarization repetitions at a submaximal inten-sity at the beginning of each repetition, and it will begin with the non-surgical ex-tremity, followed by the tests on the surgical extremity. Three effective MVIC attempts will be conducted, each lasting 5 seconds, with a 30-second rest interval between each repetition .

SECONDARY OUTCOMES:
Anterior Cruciate Ligament - Quality of Life Questionnaire (ACL - QOL) | At baseline, 30days post-surgery, 60days post-surgery, 90days post-surgery and 180days post-surgery
  This scale is of a continuous quantitative nature. It serves as a Patient-Reported Outcome Measure to assess the impact on the lives of patients with ACL, both pre- and post-treatment, regardless of whether the treatment is surgical or non-surgical. The questionnaire comprises 32 items, categorized into 5 domains: symptoms and physical prob-lems (5 items), work-related problems (4 items), sports participation/competition (12 items), lifestyle (6 items), and social and emotional aspects (5 items). Each domain is allocated a proportional score based on the number of items it contains and is evaluated using a 100-millimeter visual analog scale (VAS). A higher score indicates a better quali-ty of life for the patient. This scale was validated in Spanish, demonstrating a Cronbach's alpha of 0.81 and 0.94 and an intraclass correlation coefficient (ICC) that exhibited good consistency, ranging from 0.88 to 0.96
Lysholm Scale | At baseline, 30days post-surgery, 60days post-surgery, 90days post-surgery and 180days post-surgery
  Its purpose is to evaluate knee functionality in various types of ligament injuries, with the objective of monitoring the progression following an intervention and/or assessing knee deterioration in specific pathologies. The scale comprises eight items (limping, use of support for ambulation, instability, pain, locking, swelling, ability to ascend stairs, and ability to squat). It is evaluated on a scale of 0 - 100, with 100-95 being classified as excellent, 94-84 as good, 83-65 as fair, and less than 65 as poor. Furthermore, each item and the overall score are analysed independently. This scale demonstrates a Cronbach's alpha of 0.737 and an intraclass correlation coefficient of 0.844.
Functional Jump Test | 60days post-surgery, 90days post-surgery and 180days post-surgery
  Functional Jump Test have been commonly used for the evaluation of patients after ACLR, especially to assess the Limb Symmetry Index (LSI). Consist in 8 jump tests: Single Hop for Distance (SHD), 6m Timed Hop (6MTH), Triple Hop for Distance (THD), Triple Crossover Hop for Distance (TCHD), Single Medial Hop for Distance (MHD), Single Lateral Hop for Distance (LHD), Single Limb Countermovement Jump for Height (SLCMJ), and Timed Speedy Hop Test (TSHT)
Tampa Scale of Kinesiophobia | At baseline, 30days post-surgery, 60days post-surgery, 90days post-surgery and 180days post-surgery
  Tampa Scale of Kinesiophobia is a self-administered questionnaire composed of different questions with a 4-point Likert scale ranging from "strongly disagree" to "strongly agree.".
Pain Catastrophizing Scale | At baseline, 30days post-surgery, 60days post-surgery, 90days post-surgery and 180days post-surgery
  Pain Catastrophizing Scale (PCS) is a self-administered questionnaire (13 items on a Likert-type scale from 0 to 4), will be used in this study to assess the level of catastrophizing in the presence of pain.
EGGTMS | At baseline, 90days post-surgery, 180days post-surgery
  Brain Sight ® software to register the hotspot or point of greatest cortical activity following TMS stimulation. The hotspot helps establish the stimulation point to detect the motor threshold of activity using TMS.

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic Univerity of Valencia, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided
The data presented in this study are available on request from the corresponding author